CLINICAL TRIAL: NCT00726882
Title: A Follow-up Study to Assess the Evolution and Persistence of Resistance to ABT-333 After Discontinuation of ABT-333 Therapy in HCV Genotype-1 Infected Subjects Who Participated in Phase 1, 2, or 3 ABT-333 Clinical Studies
Brief Title: A Follow-up Assessment of Resistance to ABT-333 in Hepatitis C Virus (HCV)-Infected Subjects Who Have Received ABT-333 in ABT-333 Studies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: M10-459
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2014-12

CONDITIONS: HCV Infection
Keywords: HCV Infection
MeSH Terms: conditions — Hepatitis C | interventions — dasabuvir

ARMS (1):
- HCV-infected Participants (Other): Hepatitis C virus (HCV)-infected participants who received ABT-333 at any dose level or matching placebo in a prior clinical study involving ABT-333.
  Participants received no treatment in this follow-up study.
  Interventions: Procedure: Blood sample collection only; Drug: ABT-333

INTERVENTIONS:
Procedure: Blood sample collection only — Approximately monthly collection of blood samples.
Drug: ABT-333 — Previous treatment in prior ABT-333 studies.
  Other Names: dasabuvir

SUMMARY:
The purpose of this follow-up study is to evaluate the frequency and persistence of specific viral mutations in response to treatment with ABT-333 (dasabuvir).

DETAILED DESCRIPTION:
This Phase 2, multicenter study was conducted in HCV-infected participants who received ABT-333 at any dose level or matching placebo in a prior clinical study involving ABT-333. Hepatitis C virus (HCV)-infected participants who received ABT-333 at any dose level or matching placebo in Study M10-351 Substudy 2 (NCT00696904; ABT-333 dosing duration was 2 days) and Study M10-380 (NCT00851890; ABT-333 dosing duration was 28 days) were eligible.

After receiving at least 1 dose of ABT-333 or placebo, subjects were assessed for participation in this rollover study and asked to review the informed consent. The day of study completion or early discontinuation from the prior ABT-333 clinical study served as the baseline assessment. If it was found that a participant received placebo during the previous ABT-333 clinical study, the sites were instructed to discontinue the participant from this study.

This study included approximately monthly blood sample collection procedures for 48 weeks, and no treatment was provided during this time.

ELIGIBILITY:
Inclusion Criteria:

- Main Selection Criteria: Subject received ABT-333 or matching placebo in a prior clinical study involving ABT-333.

Exclusion Criteria:

- The investigator considers the subject unsuitable for the study for any reasons inclusive of, but not limited to, failure to comply with study procedures in prior ABT-333 clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Cohen, MD, Study Director — AbbVie
Locations (7):
- United States (6):
  - Site Reference ID/Investigator# 17665, Anaheim, California
  - Site Reference ID/Investigator# 17367, Los Angeles, California
  - Site Reference ID/Investigator# 17672, Los Angeles, California
  - Site Reference ID/Investigator# 10381, Orlando, Florida
  - Site Reference ID/Investigator# 17667, Baton Rouge, Louisiana
  - Site Reference ID/Investigator# 14461, San Antonio, Texas
- Site Reference ID/Investigator# 11141, Santurce, Puerto Rico

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hepatitis C virus (HCV)-infected participants who received ABT-333 at any dose level or matching placebo in Study M10-351 Substudy 2 (NCT00696904) or Study M10-380 (NCT00851890).
Period: Overall Study
Arm/Group | HCV-infected Participants
Started | 35
Received ABT-333 in Study M10-380 | 22 (Participants who received ABT-333 (and not placebo) in previous study (NCT00851890/M10-380).)
Received ABT-333 in Study M10-351 | 6 (Participants who received ABT-333 (and not placebo) in previous study (NCT00696904/M10-351).)
Completed | 13
Not Completed | 22
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 7
Not completed — Other | 10

BASELINE CHARACTERISTICS:
Arm/Group | HCV-infected Participants
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Persistence of Resistance-Associated Variants and Phenotypic Resistance
Description: Participants in studies M10-351 (NCT00851890) and M10-380 (NCT00696904) were analyzed for persistence of resistance-associated variants by comparing post-treatment clonal sequence data with baseline and on-treatment sequence data from M10-351 and M10-380 studies to assess amino acid changes. Phenotypic resistance to ABT-333 was assessed by calculating the fold change in half maximal effective concentration (EC50) of post-treatment samples compared with the EC50 value for the corresponding baseline sample as determined for M10-351 and M10-380 studies. The number of participants with variants at resistance-associated amino acid positions and phenotypic resistance at post-treatment time points are presented. Variants are included if the absolute percent of total clones encoding the variant was at least 10% greater than at baseline in a post-treatment sample.
Time Frame: Baseline (day of study completion or early discontinuation from the prior ABT-333 clinical study), 48 weeks
Population: Resistance analyses included all participants who received ABT-333 in the previous study who had sufficient HCV RNA recovered from samples collected during this study for genotypic and phenotypic analysis to proceed. m, n = the number of evaluable participants for the analysis specified for M10-380 and M10-351, respectively.
Measure: Number; unit: participants
Groups:
- Participants From Study M10-380: Hepatitis C virus (HCV)-infected participants who received ABT-333 at any dose level in the prior clinical study (NCT00851890/M10-380) involving ABT-333.
  Participants received no treatment in this follow-up study.
- Participants From Study M10-351: Hepatitis C virus (HCV)-infected participants who received ABT-333 at any dose level in the prior clinical study (NCT00696904/M10-351) involving ABT-333.
  Participants received no treatment in this follow-up study.
Arm/Group | Participants From Study M10-380 | Participants From Study M10-351
Number analyzed (Participants) | 5 | 4
participants
  Post-Treatment Variants in NS5B (m=5; n=3) | 4 | 0
  Post-Treatment Resistance > 10-fold (m=5; n=4) | 2 | 0

2. Secondary Outcome: Number of Participants With Serious Adverse Events Related to Study Procedures
Description: Only serious adverse events that the investigator considered causally related to study procedures (i.e., venipuncture) were to be collected in this study. A serious adverse event was defined as any untoward medical occurrence in a clinical investigation subject that the investigator believed to be causally related to a study procedure and met at least 1 of the following criteria: death, life-threatening, hospitalization or prolongation of hospitalization, congenital anomaly, persistent or significant disability/incapacity, important medical event requiring medical or surgical intervention to prevent serious outcome, elective or spontaneous abortion.
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | HCV-infected Participants
Number analyzed (Participants) | 35
participants | 0

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: Adverse events and serious adverse events (other than those related to study procedures) were not collected in this study, per protocol.
Arm/Group | HCV-infected Participants
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.